CLINICAL TRIAL: NCT05584670
Title: A Phase 1/2, Open Label, First-in-human, Dose Escalation and Expansion Study for the Evaluation of Safety, Pharmacokinetics, Pharmacodynamics, and Anti-tumor Activity of SAR445877 Administered as Monotherapy or in Combination With Other Anticancer Therapies in Adults With Advanced Solid Tumors
Brief Title: A First-in-human, Dose Escalation and Dose Expansion Study of SAR445877 in Adult Participants With Advanced Solid Tumors
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Sanofi (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: TCD17620; U1111-1277-4827 (Registry Identifier: ICTRP); 2023-507141-28 (Registry Identifier: CTIS); 2022-001239-95 (EudraCT Number)
Record Dates: First submitted 2022-10-07; First posted 2022-10-18 (Actual); Last update posted 2026-01-20 (Actual); Status verified 2026-01

CONDITIONS: Solid Tumor
MeSH Terms: interventions — Cetuximab; Bevacizumab; Nivolumab; Ipilimumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (18):
- SAR445877 Escalation Phase (Part 1A) (Experimental): SAR445877 monotherapy will be administered intravenously in participants with solid tumors over a 14-day cycle.
  Interventions: Drug: SAR445877
- SAR445877 Escalation Phase (Part1B) (Experimental): SAR445877 will be administered intravenously in combination with ADG126 in participants with advanced unresectable or metastatic melanoma, non-small cell lung cancer (NSCLC); renal cell carcinoma (RCC), hepatocellular carcinoma (HCC), colorectal cancer (MSIH/dMMR), malignant pleural mesothelioma or esophageal squamous cell carcinoma (ESCC).
  Interventions: Drug: SAR445877; Drug: ADG126
- SAR445877 Escalation Phase (Part 1C) (Experimental): SAR445877 will be administered intravenously in combination with bevacizumab in participants with metastatic colorectal cancer (CRC).
  Interventions: Drug: SAR445877; Drug: Bevacizumab
- SAR445877 Expansion/Optimization Phase: Cohort A1 (Part 2A) (Experimental): SAR445877 monotherapy will be administered intravenously (IV) in participants with non-small cell lung cancer (NSCLC).
  Interventions: Drug: SAR445877
- SAR445877 Expansion/Optimization Phase: Cohort A2 (Part 2A) (Experimental): SAR445877 monotherapy will be administered intravenously (IV) in participants with non-small cell lung cancer (NSCLC).
  Interventions: Drug: SAR445877
- SAR445877 Expansion/Optimization Phase: Cohort B (Part 2A) (Experimental): SAR445877 monotherapy will be administered intravenously in participants with hepatocellular carcinoma (HCC).
  Interventions: Drug: SAR445877
- SAR445877 Expansion/Optimization Phase: Cohort C1 (Part 2A) (Experimental): SAR445877 monotherapy will be administered intravenously in participants with gastric cancer/gastro esophageal junction adenocarcinoma (GC/GEJ).
  Interventions: Drug: SAR445877
- SAR445877 Expansion/Optimization Phase: Cohort C2 (Part 2A) (Experimental): SAR445877 monotherapy will be administered intravenously in participants with gastric cancer/gastro esophageal junction adenocarcinoma (GC/GEJ).
  Interventions: Drug: SAR445877
- SAR445877 Expansion/Optimization Phase: Cohort D (Part 2A) (Experimental): SAR445877 monotherapy will be administered intravenously IV in participants with immune infiltrated tumor type.
  Interventions: Drug: SAR445877
- SAR445877 Expansion/Optimization Phase: Cohort E1 (Part 2B) (Experimental): SAR445877 monotherapy will be administered intravenously in participants with colorectal cancer (CRC).
  Interventions: Drug: SAR445877
- SAR445877 Expansion/optimization Phase: Cohort E2 (Part 2A) (Experimental): SAR445877 monotherapy will be administered intravenously in participants with colorectal cancer (CRC).
  Interventions: Drug: SAR445877
- SAR445877 Expansion/optimization Phase: Cohort E3 (Part 2B) (Experimental): SAR445877 will be administered intravenously in combination with cetuximab in participants with colorectal cancer.
  Interventions: Drug: SAR445877; Drug: Cetuximab
- SAR445877 Japan Cohort F (Experimental): SAR445877 monotherapy will be administered intravenously in participants with advanced unresectable or metastatic solid tumor, from Japan.
  Interventions: Drug: SAR445877
- SAR445877 Expansion/Optimization Phase Cohort G1 (Part 2C) (Experimental): SAR445877 will be administered intravenously in combination with ADG126 in participants with metastatic melanoma.
  Interventions: Drug: SAR445877; Drug: ADG126
- SAR445877 Expansion/Optimization Phase Cohort G2 (Part 2C) (Experimental): SAR445877 will be administered intravenously in combination with ADG126 in participants with metastatic melanoma.
  Interventions: Drug: SAR445877; Drug: ADG126
- SAR445877 Expansion/Optimization Phase Cohort G3 (Part 2C) (Experimental): The Standard of Care (nivolumab and ipilimumab) will be administered intravenously in participants with metastatic melanoma.
  Interventions: Drug: Nivolumab; Drug: Ipilimumab
- SAR445877 Expansion/Optimization Phase Cohort H1 (Part 2D) (Experimental): SAR445877 will be administered intravenously in combination with bevacizumab in participants with advanced unresectable or metastatic CRC.
  Interventions: Drug: SAR445877; Drug: Bevacizumab
- SAR445877 Expansion/Optimization Phase Cohort H2 (Part 2D) (Experimental): SAR445877 will be administered intravenously in combination with bevacizumab in participants with advanced unresectable or metastatic CRC.
  Interventions: Drug: SAR445877; Drug: Bevacizumab

INTERVENTIONS:
Drug: SAR445877 — Concentrate for solution for infusion
  Arms: SAR445877 Escalation Phase (Part 1A); SAR445877 Escalation Phase (Part 1C); SAR445877 Escalation Phase (Part1B); SAR445877 Expansion/Optimization Phase Cohort G1 (Part 2C); SAR445877 Expansion/Optimization Phase Cohort G2 (Part 2C); SAR445877 Expansion/Optimization Phase Cohort H1 (Part 2D); SAR445877 Expansion/Optimization Phase Cohort H2 (Part 2D); SAR445877 Expansion/Optimization Phase: Cohort A1 (Part 2A); SAR445877 Expansion/Optimization Phase: Cohort A2 (Part 2A); SAR445877 Expansion/Optimization Phase: Cohort B (Part 2A); SAR445877 Expansion/Optimization Phase: Cohort C1 (Part 2A); SAR445877 Expansion/Optimization Phase: Cohort C2 (Part 2A); SAR445877 Expansion/Optimization Phase: Cohort D (Part 2A); SAR445877 Expansion/Optimization Phase: Cohort E1 (Part 2B); SAR445877 Expansion/optimization Phase: Cohort E2 (Part 2A); SAR445877 Expansion/optimization Phase: Cohort E3 (Part 2B); SAR445877 Japan Cohort F
Drug: Cetuximab — Solution for infusion
  Other Names: Erbitux
  Arms: SAR445877 Expansion/optimization Phase: Cohort E3 (Part 2B)
Drug: ADG126 — Solution for infusion
  Arms: SAR445877 Escalation Phase (Part1B); SAR445877 Expansion/Optimization Phase Cohort G1 (Part 2C); SAR445877 Expansion/Optimization Phase Cohort G2 (Part 2C)
Drug: Bevacizumab — Solution for infusion
  Other Names: bevacizumab-bvzr, Zirabev®
  Arms: SAR445877 Escalation Phase (Part 1C); SAR445877 Expansion/Optimization Phase Cohort H1 (Part 2D); SAR445877 Expansion/Optimization Phase Cohort H2 (Part 2D)
Drug: Nivolumab — Solution for infusion
  Other Names: Opdivo®
  Arms: SAR445877 Expansion/Optimization Phase Cohort G3 (Part 2C)
Drug: Ipilimumab — Solution for infusion
  Other Names: Yervoy®
  Arms: SAR445877 Expansion/Optimization Phase Cohort G3 (Part 2C)

SUMMARY:
This is a Phase 1/2, open label, multiple cohort study to assess the safety and preliminary efficacy of SAR445877 as a monotherapy or in combination with other anticancer therapies for participants aged at least 18 years with advanced unresectable or metastatic solid tumors.

The study will include 2 parts:

A dose escalation Part 1: for finding the therapeutic dose(s) of SAR445877 in a monotherapy given every 2 weeks (Q2W) or weekly (QW) and in combination with other anticancer therapies when applicable.

A multicohort dose expansion/dose optimization Part 2: for the assessment of safety and preliminary efficacy of SAR445877 in monotherapy and in combination with cetuximab or with next generation aCTLA4 (ADG126) or with bevacizumab. 2 recommended doses for expansion/optimization of SAR445877 identified from dose escalation part 1 will be tested in different indications in monotherapy and in combination with other anticancer therapies as applicable.

Approximately 542 participants will be exposed to the study intervention:

* approximately 123 participants in part 1,
* up to 410 participants in expansion/dose optimization part (part 2)
* and up to 9 participants in Japan cohort F.

DETAILED DESCRIPTION:
The duration of the study for a participant will include:

* Screening Period: up to 28 days
* Treatment Period: enrolled and exposed participants will receive continuous treatment until progressive disease (PD), or an occurrence of an unacceptable AE, a withdrawal of consent, or until other permanent discontinuation criteria described in the protocol are met.

The End of Treatment (EOT) visit will occur 30 days ±7 days from the last IMP administration or prior to the initiation of further therapy, whichever occurs first.

The follow-up period will occur until disease progression, the start of new anticancer therapy, death, or withdrawal of participant's consent, whichever comes first.

ELIGIBILITY:
Inclusion Criteria:

1. Dose escalation Part 1A and Japan Cohort F

   * Participants with advanced unresectable or metastatic solid tumors for which, in the judgement of the investigator, no standard alternative therapy is available or is not in the best interest of the participant
2. Dose escalation Part 1B

   * Participants with advanced unresectable or metastatic melanoma, NSCLC; renal cell carcinoma (RCC); HCC, colorectal cancer (MSI-H/dMMR), malignant pleural mesothelioma or esophageal squamous cell carcinoma (ESCC). and for who, in the judgement of the investigator, no standard alternative therapy is available or is not in the best interest of the participant.
3. Dose escalation Part 1C

   * Histologically or cytologically confirmed diagnosis of advanced unresectable or metastatic colorectal cancer
   * Participants with RAS-mutant and BRAF-mutant colorectal cancer are eligible for enrollment.
4. Dose expansion/optimization Part 2

   Cancer diagnosis:
   * Participants in Cohorts A1 and A2 (Part 2A): Histologically or cytologically confirmed diagnosis of metastatic non-small cell lung cancer (NSCLC)
   * Participants in Cohort B (part 2A): Histologically or cytologically confirmed diagnosis of advanced unresectable or metastatic hepatocellular carcinoma (HCC), or clinically by American Association for the Study of Liver Diseases (AASLD) criteria in cirrhotic participants (participants without cirrhosis must have had histological confirmation of diagnosis)
   * Participants in Cohorts C1 and C2 (part 2A):

     * Histologically or cytologically confirmed diagnosis of advanced unresectable or metastatic gastric cancer (GC) or Siewert Type 2 & 3 gastro esophageal junction (GEJ) adenocarcinoma
     * Disease with any CPS scoring. No need for CPS determination at local laboratory
     * Participants must have MSI (metastatic microsatellite instability) or MMR (mismatch repair) status known or determined locally and must have non-MSI-H or proficient MMR (pMMR) disease to be eligible.
     * Participants with unknown HER2/neu status must have their HER2/neu status determined locally. Participants with HER2/neu negative are eligible. Participants with HER2/neu positive tumors must have documentation of disease progression on treatment containing an approved HER2 targeted therapy to be eligible.
   * Participants in Part 2A Cohorts E1 and E2, Part 2B Cohort E3 and Part 2D Cohorts H1 and H2: Histologically or cytologically confirmed diagnosis of advanced unresectable or metastatic colorectal cancer.
   * Participants in Part 2A Cohorts E1, and E2 and Part 2B Cohort E3 MSI status:

   Participants must have MSI status known or determined locally and must have non- MSI-H disease to be eligible.
   * Participants in Part 2A Cohorts E1, E2, Part 2B Cohort E3 and Part 2D Cohorts H1 and H2: Participants with RAS-mutant and BRAF-mutant colorectal cancer are eligible for enrollment.
   * Part 2C Cohorts G1, G2 and G3: Participants with histologically confirmed unresectable locally advanced or metastatic melanoma
5. Prior anticancer therapy (For dose expansion/optimization Part 2 only)

   * Participants in Cohorts A1 and A2: Participants must have received at least 1 systemic therapy for the metastatic setting and must not be amenable to the available SOC.
   * Participants in Cohort B: Participants who have received at least 1 prior anticancer therapy, including an anti-PD1/PD-L1 containing regimen, and for whom have progressed after a primary or secondary resistance to an anti-PD1/PD-L1.
   * Participants in Cohorts C1 and C2: Participants should have failed or relapsed after at least 1 prior line of treatment which may or may not include an anti-PD1/PD-L1-based treatment depending on local standard of care.
   * Participants in Cohort D: Participants must have received at least 1 systemic therapy for their advanced/ metastatic setting and must not be amenable to the available SOC.
   * Participants in Part 2A Cohorts E1 and E2 and Part 2D Cohorts H1 and H2 should have failed or relapsed on at least 2 prior regimens.
   * Participants in cohort E3 should have failed or relapsed on at least 1 prior regimen. Participants who have received cetuximab or other anti-EGFR therapy as part of their prior line of treatment are eligible.
   * Part 2C Cohorts G1, G2 and G3: Participants must have received at least one prior line of therapy for advanced/metastatic melanoma and/or does not have any standard of care (SoC) treatment option or decline or is intolerant to be treated with SoC treatment.

Measurable Disease:

* At least 1 measurable lesion per RECIST 1.1 criteria

Part 1C and Part 2D: Adequate coagulation function for all participants. For participants receiving anti-coagulant therapy (except platelet anti-aggregates) the adequate therapeutic levels of INR should be confirmed.

Capable of giving signed informed consent.

Exclusion Criteria:

* Eastern Cooperative Oncology Group (ECOG) performance status of ≥2
* Predicted life expectancy ≤3 months
* For participants with HCC- Cohort B (Part 2): Child Pugh Class B or C liver score. Participants with Child Pugh Class B-7 score are allowed for Part 1.
* Diagnosed of any other malignancies, either progressing or requiring active treatments, within 2 years prior to enrollment
* Known active brain metastases or leptomeningeal metastases
* History of treatment-related immune-mediated (or immune-related) AEs from immune-modulatory agents (including but not limited to anti-PD1/PD-L1 agents and anti-cytotoxic T lymphocyte associated protein 4 monoclonal antibodies) that caused permanent discontinuation of the agent, or that were Grade 4 in severity or have not resolved to Grade ≤1
* Has any condition requiring ongoing/continuous corticosteroid therapy (>10 mg prednisone/day or an anti-inflammatory equivalent) within 1 week prior to the first dose of the study medicine
* Any clinically significant cardiac (including valvular) or vascular (thromboembolic disorders) disease, within 6 months prior to the first IMP administration
* Ongoing or recent (within 2 years) evidence of significant autoimmune disease that required treatment with systemic immunosuppressive treatments, which may suggest risk for immune-related adverse events
* Has a known history or any evidence of interstitial lung disease or active, non-infectious pneumonitis within 3 years prior to the first dose of the study drug.
* Organ transplant requiring immunosuppressive treatment
* Uncontrolled or active infection with human immunodeficiency virus (HIV), hepatitis B, or hepatitis C infection, or has a diagnosis of immunodeficiency

NOTE: Other Inclusion/Exclusion criteria may apply.

The above information is not intended to contain all considerations relevant to a potential participation in a clinical trial.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 542 (Estimated)
Dates: Start 2022-11-29 (Actual); Primary Completion 2027-01-19 (Estimated); Study Completion 2028-06-28 (Estimated)

PRIMARY OUTCOMES:
Dose escalation part 1A, 1C and Japan Cohort F: Presence of dose-limiting toxicities (DLTs) in Cycles 1 and 2 | Cycles 1 & 2 - 14 days per cycle
  DLTs will be defined using NCI CTCAE version 5.0 or ASTCT criteria for CRS or immune effector cell-associated neurotoxicity syndrome (ICANS)
Dose escalation part 1B: Presence of dose-limiting toxicities (DLTs) in Cycle 1 to 3 in part B | Cycle 1 to 3 -14 days per cycle
Dose escalation and Japan Cohort F: Percentage of participants experiencing treatment-emergent adverse events (TEAEs) | The time from the first dose of study interventions up to 30 days after last dose of study interventions
  Presence of TEAEs, SAEs, and lab abnormalities, according to the National Cancer Institute (NCI) Common Terminology Criteria for Adverse Events (CTCAE) Version 5.0 and American Society for Transplantation and Cellular Therapy (ASTCT) consensus grading
Dose expansion/optimization: Objective response rate (ORR) | From baseline to the end of dose expansion/optimization (up to 2 years)
  Proportion of participants who have a confirmed complete response (CR) or a partial response (PR), as the best overall response (BOR) determined by the Investigator as per the Response Evaluation Criteria in Solid Tumors (RECIST) v1.1

SECONDARY OUTCOMES:
Dose escalation and Japan Cohort F: Objective response rate (ORR) | From baseline to the end of dose escalation (up to 2 years)
  Proportion of participants who have a confirmed complete response (CR) or a partial response (PR), as the best overall response (BOR) determined by the Investigator as per the Response Evaluation Criteria in Solid Tumors (RECIST) v1.1
Dose escalation, expansion/optimization and Japan Cohort F: Duration of response (DoR) | From baseline to the end of study (up to 2 years)
  DoR is defined as the time from first documented evidence of confirmed CR or PR until progressive disease (PD) determined by Investigator per RECIST 1.1 or death from any cause, whichever occurs first
Dose escalation, expansion/optimization and Japan Cohort F: Assessment of SAR445877 Cmax | Cycle 1 Day 1 to Day 8 or Day 14 (cycle duration of 14 days)
  Maximum plasma concentration observed
Dose escalation, expansion/optimization and Japan Cohort F: Assessment of SAR445877 AUCtau | Cycle 1 Day 1 to Day 8 or Day 14 (cycle duration of 14 days)
  Area under the concentration versus time curve calculated using the trapezoidal method during a dosing interval (T)
Dose escalation, expansion/optimization and Japan Cohort F: Assessment of SAR445877 Tmax | Cycle 1 Day 1 to Day 8 or Day 14 (cycle duration of 14 days)
  First time to reach Cmax
Dose escalation, expansion/optimization in Combination: Assessment of combined therapies Ctrough | Day 1 of each cycle to cycle 4 (cycle duration of 14 days)
Dose escalation, expansion/optimization and Japan Cohort F: Percentage of participants with presence of anti-drug antibodies (ADAs) against SAR445877 | From the first dose of Cycle 1 to 30 days after last dose of study interventions (cycle duration of 14 days)
Dose escalation, expansion/optimization: Percentage of participants with presence of anti-drug antibodies (ADAs) against ADG126 | From the first dose of Cycle 1 to 30 days after last dose of study interventions (cycle duration of 14 days)
Dose expansion/optimization: Time to response | From baseline to end of dose expansion/optimization (up to 2 years)
  Time to response is defined as the time from the first administration of investigational medicinal product (IMP) to the first documented evidence of confirmed PR or CR determined by Investigator per RECIST 1.1
Dose expansion/optimization: Clinical Benefit Rate | From baseline to end of dose expansion/optimization (up to 2 years)
  Clinical Benefit Rate including confirmed CR or PR at any time or stable disease (SD) of at least 6 months determined by Investigator per RECIST 1.1
Dose expansion/optimization: Progression-free survival | From baseline to end of dose expansion/optimization (up to 2 years)
  PFS is defined as the time from the date of first administration of IMP to the date of the first documented disease progression determined by Investigator as per RECIST 1.1 or death from any cause, whichever occurs first
Dose expansion/optimization: Overall survival | From baseline to end of dose expansion/optimization (up to 2 years)
  Overall survival (OS) is defined as the time from the first dose of IMP to the date of death due to any cause.
Dose expansion/optimization: Number of participants with Adverse events (AE) | The time from the first dose of study interventions up to 30 days after last dose of study interventions.
  Presence of adverse events (AEs) graded according to the National Cancer Institute (NCI) Common Terminology Criteria for Adverse Events (CTCAE) Version 5.0 or American Society for Transplantation and Cellular Therapy (ASTCT) consensus grading

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Sciences & Operations, Study Director — Sanofi
Locations (22):
- United States (9):
  - Christiana Care Health System- Site Number : 8400011, Newark, Delaware
  - University of Iowa- Site Number : 8400014, Iowa City, Iowa
  - University of Kansas Cancer Center Clinical Research Center (Fairway) Site Number : 8400008, Fairway, Kansas
  - Barbara Ann Karmanos Cancer Institute - Detroit- Site Number : 8400006, Detroit, Michigan
  - John Theurer Cancer Center Site Number : 8400001, Hackensack, New Jersey
  - NYU Langone Medical Center-New York- 550 1st Ave - BRANY - PPDS- Site Number : 8400013, New York, New York
  - Rhode Island Hospital Site Number : 8400004, Providence, Rhode Island
  - University of Texas MD Anderson Cancer Center Site Number : 8400005, Houston, Texas
  - Fred Hutchinson Cancer Center - 825 Eastlake Ave E- Site Number : 8400010, Seattle, Washington
- Chile (4):
  - Servicios Médicos URUMED SpA_Investigational Site Number : 1520002, Rancagua, General Bernardo O'Higgins
  - BIOCINETIC Ltda_Investigational Site Number : 1520008, Santiago, Reg Metropolitana de Santiago
  - Fundacion Arturo Lopez Perez (FALP) - Providencia - Jose Manuel Infante 805_Investigational Site Number : 1520007, Providencia
  - Centro de Investigacion Clinica Bradford Hill_Investigational Site Number : 1520004, Recoleta
- Israel (4):
  - Hadassah Medical Center - PPDS_Investigational Site Number : 3760005, Jerusalem, Jerusalem
  - Shamir Medical Center_Investigational Site Number : 3760004, Be’er Ya‘aqov
  - Sheba Medical Center - PPDS_Investigational Site Number : 3760003, Ramat Gan
  - Tel Aviv Sourasky Medical Center Ichilov - PPDS_Investigational Site Number : 3760001, Tel Aviv
- Investigational Site Number : 3920001, Kashiwa-Shi, Japan
- Netherlands (2):
  - Het Nederlands Kanker Instituut Antoni Van Leeuwenhoek Ziekenhuis_Investigational Site Number : 5280001, Amsterdam, North Holland
  - Erasmus MC_Investigational Site Number : 5280003, Rotterdam, South Holland
- Spain (2):
  - Instituto de Investigacion Oncologica Vall d'Hebron (VHIO) - EPON_Investigational Site Number : 7240007, Barcelona
  - START MADRID_Hospital Universitario HM Sanchinarro - CIOCC_Investigational Site Number : 7240005, Madrid

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers may request access to patient level data and related study documents including the clinical study report, study protocol with any amendments, blank case report form, statistical analysis plan, and dataset specifications. Patient level data will be anonymized, and study documents will be redacted to protect the privacy of trial participants. Further details on Sanofi's data sharing criteria, eligible studies, and process for requesting access can be found at: https://vivli.org

REFERENCES:
- See also: TCD17620 Plain Language Results Summary — https://www.trialsummaries.com/Study/StudyDetails?id=25350&tenant=MT_SNY_9011